CLINICAL TRIAL: NCT01453959
Title: Fludrocortisone's Test in the Identification of Salt Sensitivity
Brief Title: Fludrocortisone's Test in Salt Sensitivity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Decio Mion Jr., Clinical Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPESP 2010/170726
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension
Keywords: hypertension; salt sensitivity; fludrocortisone
MeSH Terms: conditions — Hypertension | interventions — Fludrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet cycles (Other): The patient will be analysed for salt sensitivity by two cycle of diets: low salt diet(40mEq Sodium/day by 7 days) and high salt diet (240mEq Sodium/day by 7 days). After 4 weeks without any intervention, the patient will received fludrocortisone in a dose of 0.4 mg/day for 7 days.
  Interventions: Other: Diet cycles
- Fludrocortisone (Other): The patient will received fludrocortisone in a dose of 0.4 mg/day for 7 days. After 4 weeks without any intervention, the patient will be analysed for salt sensitivity by two cycle of diets: low salt diet(40mEq Sodium/day by 7 days) and high salt diet (240mEq Sodium/day by 7 days).
  Interventions: Drug: Fludrocortisone

INTERVENTIONS:
Drug: Fludrocortisone — Fludrocortisone in a dose of 0.4 mg/day for 7 days
  Arms: Fludrocortisone
Other: Diet cycles — Two cycle of diets: low salt diet(40mEq Sodium/day by 7 days) and high salt diet (240mEq Sodium/day by 7 days)
  Arms: Diet cycles

SUMMARY:
The main hypothesis of this study is look for a clinical and fast test to identify salt sensitivity by administration of fludrocortisone.

DETAILED DESCRIPTION:
The relationship between excessive salt intake and hypertension is well established in the literature. However, the intensity of blood pressure increase in response to such intake varies among individuals. The salt sensitivity is, therefore, measurement of blood pressure response to the variation of salt content in the diet in each individual. The importance of sensitivity to salt has been well demonstrated, with higher mortality in both hypertensive patients and in normotensives subjects. Despite this importance, the methods of assessment salt sensitivity are difficult to be adopted into clinical practice. The test considered the standard for sensitivity to salt is the administration of two cycles of low and high sodium diets, and checked the change in mean arterial pressure between the end of the first and second cycles. Note, therefore, that the supply of diets, as well as patient compliance, are difficult in routine clinical practice. The aim of this study is to compare the administration of fludrocortisone in identifying patients with salt sensitive with the gold standard low and high sodium diets. A experimental cross-over study, with 40 uncomplicated hypertensive patients, will be conducted. Initially, all patients are going to stay in a period of washout of antihypertensive medications with a duration of four weeks, receiving placebo. Following this, they will be submitted for salt sensitivity in two phases: during the cycle of diets, lasting two weeks, and during administration of fludrocortisone in a dose of 0.4 mg/day for 7 days. Between these two phases will be a period of four weeks. The order of the phases will be divided by simple randomization. Moreover, we will evaluate the relationship between blood pressure and 24-hour urinary sodium excretion during cycles of diet low / high sodium. After the study, the test accuracy of fludrocortisone will be analyzed by calculating the sensitivity, specificity and positive predictive value and negative, in addition to the construction of a ROC curve for determining a cutoff point to improve the specificity and sensitivity of the test.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 65 years
* Both sexes and all ethnicities;
* Body Mass Index (BMI) between 20 and 30 kg/m2;
* Patients with hypertension with systolic blood pressure (SBP) between 140 and 159 mmHg and diastolic blood pressure (DBP) between 90 mm Hg and 99 mm Hg, without medication or after four weeks of placebo

Exclusion Criteria:

* Moderate/severe hypertension (BP ≥ 160/100 mm Hg) or secondary cause of hypertension;
* Use of more than two antihypertensive classes at the time of selection;
* Presence of diabetes mellitus or other endocrine disorders;
* Presence of renal impairment (creatinine clearance <60 ml / min, calculated by Cockcroft-Gault formula);
* Presence of heart failure;
* Presence of cardiac arrhythmias;
* History of stroke, coronary heart disease (myocardial infarction, angina) and peripheral vascular insufficiency;
* Presence of liver failure;
* Alcoholism;
* Psychiatric disorders;
* Use of anovulatory or continuous use of other drugs, such as hormonal or nonhormonal anti-inflammatory drugs that may interfere with blood pressure.
* Pregnant women

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-09 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure difference | Baseline and 11 weeks
  Patient will be analised for salt sensitivity in two phases: during the cycle of diets (low and high salt), lasting two weeks, and during administration of fludrocortisone (0.4 mg/day for 7 days). In the begin and finish of each phase (diets and fludrocortisone), blood pressure will be measure by oscilometric methods in the office and by ambulatory blood pressure monitoring (ABPM) and home blood pressure monitoring (HBPM) out-of-office. The difference of blood pressure between each phase will be used to classify the patient in salt sensitive or salt resistant.

CONTACTS AND LOCATIONS:
Overall Officials: Decio Mion Junior, MD, PhD, Principal Investigator — General Hospital of School of Medicine - Universiy of Sao Paulo
Locations (1):
- General Hospital of School of Medicine - Universiy of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Pio-Abreu A, de Castro I, da Silva GV, Ortega KC, Mion D Jr. Oral Fludrocortisone Test for Salt-Sensitive Screening in Hypertensive Patients: A Randomized Crossover Trial. Int J Hypertens. 2018 Nov 15;2018:7437858. doi: 10.1155/2018/7437858. eCollection 2018. PMID 30581606